CLINICAL TRIAL: NCT00900419
Title: Biomarkers and Dysplastic Respiratory Epithelium
Brief Title: Biomarkers in Patients With Respiratory Tract Dysplasia or Lung Cancer, Head and Neck Cancer, or Aerodigestive Tract Cancer and in Normal Volunteers
Status: Recruiting | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 00-1108.cc; SPORE 24 (Other: SPORE Number); P50CA058187 (NIH)
Record Dates: First submitted 2009-05-09; First posted 2009-05-12 (Estimated); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Esophageal Cancer; Head and Neck Cancer; Lung Cancer; Precancerous Condition
Keywords: non-small cell lung cancer; small cell lung cancer; squamous lung dysplasia; hypopharyngeal cancer; laryngeal cancer; lip and oral cavity cancer; metastatic squamous neck cancer with occult primary; nasopharyngeal cancer; oropharyngeal cancer; paranasal sinus and nasal cavity cancer; salivary gland cancer; esophageal cancer; pulmonary carcinoid tumor; tongue cancer
MeSH Terms: conditions — Esophageal Neoplasms; Head and Neck Neoplasms; Lung Neoplasms; Precancerous Conditions; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Hypopharyngeal Neoplasms; Laryngeal Neoplasms; Mouth Neoplasms; Nasopharyngeal Neoplasms; Oropharyngeal Neoplasms; Salivary Gland Neoplasms; Tongue Neoplasms | interventions — Immunohistochemistry; Biopsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Sputum sample, Endobronchial biopsy, bronchial secretions, pulmonary lavage, blood and urine.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: immunohistochemistry staining method — Laboratory test
Other: laboratory biomarker analysis — Laboratory Test
Other: sputum cytology — Laboratory Test
Procedure: biopsy — Laboratory Test

SUMMARY:
RATIONALE: Studying samples of sputum and tissue in the laboratory from patients with dysplasia or cancer may help doctors identify and learn more about biomarkers related to cancer. It may also help the study of cancer in the future.

PURPOSE: This laboratory study is looking at biomarkers in patients with respiratory tract dysplasia or lung cancer, head and neck cancer, or aerodigestive tract cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine intermediate biomarkers of premalignant respiratory epithelial lesions, such as genetic mutations or altered growth factor expression, in patients with dysplasia of the respiratory epithelium or lung cancer, head and neck cancer, or aerodigestive tract cancer.

Secondary

* Establish a tissue repository of normal and dysplastic respiratory epithelium from endobronchial forceps and brush biopsy tissue from these patients and from normal volunteers.

OUTLINE: Patients are stratified according to presence of extensive and severe dysplasia of the respiratory epithelium (yes vs no).

Participants undergo sputum cytology, white-light (with or without fluorescence) bronchoscopy, and endobronchial biopsies. Participants also undergo endobronchial brushings and bronchial secretion collection and possibly bronchoalveolar lavage. Collected samples are processed by hematoxylin, eosin, and immunohistochemical staining and analyzed for specific biomarkers. Unused samples are stored in the tissue bank.

PROJECTED ACCRUAL: A total of 330 participants will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of extensive and severe dysplasia of the respiratory epithelium
* Those without dysplasia of the respiratory epithelium

  * Recruited from the SPORE Tissue Procurement Screening Project or by private or academic physicians (for patients with moderate or severe dysplasia)
* Survived 1 or more aerodigestive system carcinoma for ≥ 1 year
* Completely resected stage I non-small cell cancer
* Undergoing any of the following procedures:

  * Routine panendoscopy for patients with head and neck cancer
  * Resection of a bronchogenic carcinoma
  * Bronchoscopy for diagnosis or staging of suspected lung cancer
  * Subsequent bronchoscopy for surveillance or monitoring of response to endobronchial treatment in patients with prior high-grade dysplasia or worse
  * No asthma
  * No lung disease
  * No respiratory illness within the past 2 weeks Patients suspected of or at risk for neoplastic lung disease who are undergoing a bronchoscopy in which differential diagnostic considerations may include multiple other etiologies such as infection and other processes.
  * Patients without dysplasia will be: patients undergoing clinically indicated bronchoscopy for conditions other than suspected lung cancer.

PATIENT CHARACTERISTICS:

* No clinically apparent bleeding diathesis
* No known bleeding disorder
* No anginal
* No clinically active coronary artery disease
* No multifocal premature ventricular contractions
* No poorly controlled congestive heart failure
* No myocardial infarction within the past 6 weeks
* No cardiac dysrhythmia that is potentially life threatening
* Well-controlled atrial fibrillation or rare (< 2/min) premature ventricular contractions allowed
* No ventricular tachycardia or supraventricular tachycardia with a rapid ventricular response
* No other serious medical condition that would preclude a patient from undergoing a bronchoscopy
* No acute bronchitis or pneumonia within the past 8 weeks except when clinically proven as a possible result of lung cancer
* No hypoxemia (i.e., < 90% saturation with supplemental oxygen) before bronchoscopy

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: High Risk for Lung Cancer, suspected lung cancer, lung cancer.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2001-05-03 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Genetic mutations or altered growth factor expression | After study has completed

SECONDARY OUTCOMES:
Establishment of a tissue repository of normal and dysplastic respiratory epithelium | After study has closed

CONTACTS AND LOCATIONS:
Overall Officials: York E. Miller, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Cancer Center at UC Health Sciences Center, Aurora, Colorado, United States